CLINICAL TRIAL: NCT02866175
Title: Evaluation of the Safety and Efficacy of an Edoxaban-based Compared to a Vitamin K Antagonist-based Antithrombotic Regimen in Subjects With Atrial Fibrillation Following Successful Percutaneous Coronary Intervention (PCI) With Stent Placement.
Brief Title: Edoxaban Treatment Versus Vitamin K Antagonist in Patients With Atrial Fibrillation Undergoing Percutaneous Coronary Intervention
Acronym: ENTRUST-AF-PCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSE-EDO-01-15-EU; 2016-002683-14 (EudraCT Number)
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
Keywords: percutaneous intervention; vitamin K antagonist
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Edoxaban Regimen (Experimental): Participants will be randomized to receive edoxaban 60 mg once-daily or 30 mg once-daily and clopidogrel 75 mg once-daily (or in the presence of a documented clinical need prasugrel [5 mg or 10 mg once-daily] or ticagrelor [90 mg twice-daily] may be used) used.
  Interventions: Drug: Edoxaban; Drug: Clopidogrel; Drug: Prasugrel; Drug: Ticagrelor
- Vitamin K Antagonist Regimen (Active Comparator): Participants will be randomized to receive VKA in combination with clopidogrel 75 mg once-daily (or in the presence of a documented clinical need prasugrel [5mg or 10 mg once-daily] or ticagrelor [90 mg twice-daily] may be used) and aspirin (100 mg once-daily, for a minimum of 1 month and up to 12 months duration.
  Interventions: Drug: Clopidogrel; Drug: Prasugrel; Drug: Ticagrelor; Drug: Vitamin K antagonist

INTERVENTIONS:
Drug: Edoxaban — Edoxaban 60 mg once-daily or 30 mg once-daily in selected subjects
  Other Names: Savaysa
  Arms: Edoxaban Regimen
Drug: Clopidogrel — Clopidogrel 75 mg once-daily
  Other Names: Plavix
Drug: Prasugrel — prasugrel 5mg or 10 mg once-daily
  Other Names: Effient
Drug: Ticagrelor — ticagrelor 90 mg twice-daily
Drug: Vitamin K antagonist — VKA once-daily dosing for target international normalized ratio between 2.0 and 3.0, inclusive
  Arms: Vitamin K Antagonist Regimen

SUMMARY:
There are insufficient data on the safety and efficacy of edoxaban plus antiplatelet therapy in subjects with atrial fibrillation (AF) following percutaneous intervention (PCI) with stenting. This study is designed to evaluate the safety and to explore the efficacy of an edoxaban-based antithrombotic regimen versus a vitamin K antagonist (VKA)-based antithrombotic regimen in subjects with AF following PCI with stent placement. Bleeding is a central safety outcome in cardiovascular clinical trials, especially for antithrombotic strategies and invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Oral anticoagulant (OAC) indication for atrial fibrillation for a period of at least 12 months following successful PCI with stenting.

Eligibility is assessed 4 hours after sheath removal and within 5 days after successful PCI with stent placement. If a staged PCI is planned, eligibility is assessed after completion of the last stage.

Successful PCI definition:

The success of a PCI procedure is defined by 2 interrelated components: angiographic findings, procedural / clinical outcomes as detailed below:

Angiographic Success A minimum stenosis diameter of < 20% (as visually assessed by angiography - residual blockage or stenosis reduced to less than 20% of the artery's diameter).

Sufficient enlargement of the lumen at the target site to improve coronary artery blood flow with final thrombolysis in myocardial infarction (TIMI) flow grade 3 (visually assessed by angiography), without occlusion of a significant side branch, flow-limiting dissection, distal embolization, or angiographic thrombus.

Procedural Success No major in-hospital clinical complications(e.g. ongoing International Society on Thrombosis and Haemostasis [ISTH] major or clinical relevant non-major procedural bleeding at the time of randomization, stroke, emergency coronary artery bypass graft [CABG]).

In summary, a clinically successful PCI requires both anatomic and procedural success along with relief of signs and/or symptoms of myocardial ischemia at the time of randomization.

Exclusion Criteria:

* Bleeding risks or systemic conditions
* Known bleeding diathesis, including but not limited to,

  1. Uncontrolled active bleeding, encompassing both ISTH major and clinically relevant non-major bleeding, preceding randomization.

     Lesion or condition, if considered to be a significant risk for major bleeding. This may include but is not limited to: unresolved gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding (e.g. malignancies with metastasis), recent unresolved brain or spinal injury, recent brain, spinal or ophthalmic surgery, any intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms (of more than 3.5 cm) or major intraspinal or intracerebral vascular abnormalities.
  2. Medication-related
* International normalized ratio (INR) > 2.5 (the participant can be reconsidered at a later time, but within 5 days of sheath removal).
* Contraindication to edoxaban, VKA, acetylsalicylic acid (ASA) and/or P2Y12 antagonists;
* Concomitant treatment with other antithrombotic agents, fibrinolytic therapy and chronic nonsteroidal anti-inflammatory drugs (NSAIDs).

Concomitant conditions and therapies

* Critically ill or hemodynamically unstable subjects (at the time of randomization) including:

  1. cardiogenic shock or acute decompensated heart failure, with the requirement for vasopressor agents or inotropic support or mechanical support to support circulation
  2. respiratory failure requiring endotracheal intubation and mechanical ventilation.
* Any prior mechanical valvular prosthesis;
* Planned coronary or vascular intervention or major surgery within 12 months; Randomization must be deferred to the last stage in a multistep, multivessel PCI procedure;
* Moderate or severe mitral stenosis;
* Ischemic stroke within 2 weeks prior to randomization;
* Uncontrolled severe hypertension with a systolic blood pressure (BP) ≥180 mmHg and/or diastolic BP ≥ 120 mmHg;
* End stage renal disease (ESRD) (CrCL < 15 mL/min or on dialysis);
* Known abnormal liver function prior to randomization (including hepatic disease or biochemical evidence of significant liver derangement known prior to randomization).

Other exclusion criteria

* Any of the following abnormal local laboratory results prior to randomization:

  1. Platelet count < 50 x10^9/L
  2. Hemoglobin < 8 mg/dL
* Unable to provide written Informed Consent;
* Female participants of childbearing potential without using highly effective contraception (female of childbearing potential is defined as one who has not been postmenopausal for at least one year, or has not been surgically sterilised, or has not had a hysterectomy at least three months prior to the start of this study). Females taking oral contraceptives should have been on therapy for at least three months. Adequate contraceptives include: Combined (estrogen and progestogen containing) oral, intravaginal, transdermal, hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence;
* Pregnant or breast-feeding participants;
* Assessment that the participant is not likely to comply with the study procedures or have complete follow-up;
* Participating in another clinical trial that potentially interferes with the current study;
* Previous randomization in this study;
* Active on prescription drug abuse and addiction; abuse of illicit substances (i.e. marijuana, cocaine, methamphetamine, heroin) and alcohol abuses during the last 12 months according to the judgement of the investigator;
* Life expectancy < 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1506 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Vranckx, MD, Study Chair — Hartcentrum Hasselt; Andreas Gotte, Prof., MD, Study Chair — Medizinische Klinik II
Locations (200):
- Austria (4):
  - Medizinische Universitaetsklinik Graz, Graz
  - University Hospital Innsbruck, Innsbruck
  - Krankenhaus Hietzing, Vienna
  - Wilhelminenspital, Vienna
- Belgium (7):
  - ASZ Aalst, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - AZ St Jan, Bruges
  - Hopital Erasme, Brussels
  - University Hospital Antwerp, Edegem
  - Virga Jesse Jessa hospital, Hasselt
  - AZ Delta, Roeselare
- France (10):
  - University Hospital of Angers, Angers
  - Hopital Cote Basque, Bayonne
  - Chru Jean Minjoz, Besançon
  - Metropole Savoie Hospital, Chambéry
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hospital Henri Mondor, Créteil
  - CHU de Nice, Nice
  - Hôpital Bichat - Claude Bernard, Paris
  - Hôpital Rangueil, Service Cancérologie, Toulouse
  - Clinique Vauban, Valenciennes
- Germany (31):
  - University Hospital Aachen, Aachen
  - Universitäts-Herzzentrum Freiburg • Bad Krozingen, Bad Krozingen
  - Kerckhoff Klinik, Bad Nauheim
  - Vivantes Klinikum im Friedrichshaim, Berlin
  - Charité Benjamin Franklin, Berlin
  - Charité, Campus Virchow-Klinikum - Medizinische Klinik mit Schwerpunkt Kardiologie, Berlin
  - Staedtische Kliniken Bielefeld, Bielefeld
  - GFO Kliniken Bonn - St.-Marien-Hospital, Bonn
  - Universitätsklinikum Bonn - Medizinische Klinik II - Innere Medizin (Kardiologie, Angiologie und Pneumologie), Bonn
  - Klinikum Coburg Med. Klinik Kardiologie, Angiologie, Pneumologie, Coburg
  - St. Johannes- Hospital, Dortmund
  - Heinrich-Heine-Universität Düsseldorf - Universitätsklinikum Düsseldorf (UKD) Klinik für Kardiologie, Pneumologie und Angiologie, Düsseldorf
  - Universitaetsklinikum Freiburg Klinik für Kardiologie und Angiologie I, Freiburg im Breisgau
  - Universitäres Herzzentrum Hamburg GmbH (UHZ), Hamburg
  - Universitätsklinikum Heidelberg Klinik für Kardiologie, Angiologie und Pneumologie (Innere Medizin III), Heidelberg
  - Universitätsklinikum des Saarlandes Innere Medizin III - Kardiologie, Angiologie und internistische Intensivmedizin, Homburg
  - Universitätsklinikum Jena Klinik für Innere Medizin I, Kardiologie, Angiologie, Pneumologie, Internistische Intensivmedizin, Jena
  - Herzzentrum Leipzig - Universitätsklinik Klinik für Innere Medizin/Kardiologie, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen
  - Städtisches Klinikum Lüneburg, Lüneburg
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinik Dr. Müller GmbH & Co. KG, Peter Osypka Herzzentrum, München
  - Universitätsklinikum Münster - Department für Kardiologie und Angiologie, Münster
  - St. Vincenz-Krankenhaus Paderborn - Medizinische Klinik II, Paderborn
  - Universitätsmedizin Rostock, Rostock
  - Universitäts Klinikum Tübingen, Tübingen
  - Herzklinik Ulm, Ulm
  - Universitätsklinik Ulm - Zentrum für Innere Medizin - Klinik für Innere Medizin II, Ulm
  - Schwarzwald-Baar Klinikum - Kliniken Villingen-Schwenningen - Innere Medizin III: Kardiologie und Intensivmedizin, Villingen-Schwenningen
  - St. Josefs-Hospital - Medizinische Klinik I, Kardiologie, Wiesbaden
  - HELIOS Klinikum Wuppertal - Herzzentrum, Wuppertal
- Hungary (12):
  - Állami Szívkórház, Balatonfüred
  - Budai Irgalmasrendi Kht., Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Békés Megyei Központi Kórház, Gyula
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Jósa András Oktatókórház, Nyíregyháza
  - Pécsi Tudományegyetem, Pécs
  - Szegedi Tudományegyetem, Szeged
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár
- Italy (22):
  - Ospedale San Donato- ASL 8 Arezzo, Arezzo
  - Policlinico di Bari, Bari
  - Ospedale Maggiore C.A. Pizzardi -OR - Laboratorio di Cardiologia Interventistica, Bologna
  - AOU Materdomini, Magna Graecia University, Catanzaro
  - ASL2 Chieti - SS Maria Annunziata, Chieti
  - A.S.O.S. Croce e Carle Cuneo, Cuneo
  - AOU Sant'Anna, Ferrara
  - Ospedale Careggi, Florence
  - Ospedali Riuniti di Foggia, Foggia
  - Ospedale Alessandro Manzoni-Azienda Ospedaliera di Lecco, Lecco
  - Asst Fatebenefratelli-Sacco, Milan
  - AOU Policlinico di Modena, Modena
  - University Hospital Federico II, Napoli
  - Padova University Hospital, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Ospedale degli Infermi, Rimini
  - Ospedale degli Infermi di Rivoli, Rivoli
  - Policlinico Agostino Gemelli, Roma
  - S.Camillo Forlanini - Ospedale S.Camillo Reparto di Emodinamica, Rome
  - Bolognini Hospital Seriate, Seriate
  - "Santa Maria" University Hospital - Azienda Ospedaliera Santa Maria Di Terni, Terni
  - U.O. Cardiologia Ospedale Borgo Trento, Verona
- Lithuania (4):
  - Lithuanian University of Health Sciences hospital, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
  - Republican Siauliai Hospital, Šiauliai
  - Vilnius University Hospital "Santariskiu Clinic", Vilnius
- Netherlands (4):
  - St Antonius Hospital, Nieuwegein
  - Radboud university medical center, Nijmegen
  - Maasstad Hospital, Rotterdam
  - MC Haaglanden, The Hague
- Poland (11):
  - II Oddział Kardiologiczny, Polsko-Amerykanskie Kliniki Serca, Bielsko-Biala
  - MCSN AHoP, Chrzanów
  - III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii Polsko-Amerykanskie Kliniki Serca, Dąbrowa Górnicza
  - AHP IV DEP K-Kozle, Kędzierzyn-Koźle
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Oddział Kliniczny Kardiologii Interwencyjnej z Pododdziałem Intenyswengo Nadzoru Kardiologicznego, Krakow
  - Nzoz Salus, Lodz
  - Nyskie Centrum Sercowo-Naczyniowe, Polsko-Amerykanskie Kliniki Serca, Nysa
  - Clin-Medica OMC sp. z o.o. s.k., Skierniewice
  - X Oddział Kardiologii Inwazyjnej, Elektrofizjologii i Elektrostymulacji Polsko-Amerykanskie Kliniki Serca, Tychy
  - Instytut Kardiologii im. Prymasa Tysiaclecia Kardynala Stefana Wyszynskiego, Klinika Choroby Wieńcowej i Strukturalnych Chorób Serca, Warsaw
  - Instytut Kardiologii im. Prymasa Tysiąclecia Stefana Kardynała Wyszyńskiego; Klinika Kardiologii i Angiologii Interwencyjnej, Warsaw
- Portugal (6):
  - Hospital Garcia de Orta, EPE, Almada
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Centro Hospitalar e Universitário de Coimbra, EPE - Hospital dos Covões, Coimbra
  - Centro Hospitalar de Lisboa Central, EPE - Hospital Santa Marta, Lisbon
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
- Romania (7):
  - Emergency County Hospital Baia Mare, Baia Mare
  - "Prof. C.C. Iliescu" Emergency Institute for Cardiovascular Diseases, Bucharest
  - University Hospital of Bucharest, Bucharest
  - Saint John Emergency Hospital, Bucharest
  - Oradea Emergency County Clinical Hospital, Oradea
  - Emergency Institute of Cardiovascular Diseases and Transplantation, Târgu Mureş
  - Institutul de Boli Cardiovasculare Timisoara, Timișoara
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center -Zvezdara, Belgrade
  - Institute of CV Diseases Clinical Center of Serbia, Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- South Korea (16):
  - Pusan National University Hospital, Busan
  - Daegu Catholic University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Inje Univ. Ilsan Paik Hospital, Gyeonggi-do
  - The Catholic University of Korea St.Vincent's Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Centre, Seoul
  - SEOUL St.Maria, Seoul
  - Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Anam Hospital, Seoul
- Spain (16):
  - General University Hospital of Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Complejo Hospitalario Universitario de Granada, Granada
  - Bellvitge University Hospital, L'Hospitalet de Llobregat
  - Complejo Asistencial Universitario de León, León
  - Hospital Ramon y Cajal, Madrid
  - Clinica Universitaria San Carlos, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Álvaro Cunqueiro, Vigo
- Switzerland (2):
  - HFR Freiburg - Kantonsspital Kardiologie, Fribourg
  - Cardiocentro Ticino, Lugano
- Taiwan (10):
  - Hsinchu Mackay Memorial Hospital (HMMH), Hsinchu
  - Kaohsiung medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital (FEMH), New Taipei City
  - China Medical University Hospital (CMUH), Taichung
  - Chi-Mei Medical Center (CMMC), Tainan
  - National Cheng Kung University Hospital, Tainan
  - Cheng Hsin General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Taoyuan District
- Ukraine (27):
  - Cherkasy regional cardiological center, Cherkasy
  - Chernihiv City Hospital #2, Chernihiv
  - Chernivtsi Regional Clinical Cardiology Dispensary, Chernivtsi
  - Communal Institution Dnepropetrovsk Regional Diagnostic Center, Dnipro
  - CI "Dnipropetrovsk Joint Emergency Hospital", Dnipropetrovsk
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Kharkiv Railway Clinical Hospital N1 of Brance "Health Center" of the Public joint stock company "Ukrainian Railway", Kharkiv
  - L.T. Malaya Therapy National Institute of the National Academy of medical science of Ukraine, Kharkiv
  - Communal Health Care Institution "Regional Clinical Hospital - Center of Emergency Medical Care and Disaster Medicine", Kharkiv
  - Kharkiv City Clinical Hospital #8, Kharkiv
  - Khmelnytskyy regional hospital, Khmelnytskyi
  - Insititute of Heart of MoH Ukraine, Kyiv
  - Kyiv City Clinical Hospital#5, Kyiv
  - State Institution 'National Scientific Central Institute of Cardiology named after MD Strazhesko', Kyiv
  - Kyiv City Clinical Hospital 4, Kyiv
  - Oleksandrivska Kiyv City Clinical Hospital, Kyiv
  - Communal Institution of Kyiv Regional Rada, Kyiv
  - Lutsk City Hospital, Lutsk
  - Lviv Regional State Clinical Treatment and Diagnostic Cardiology Center, Lviv
  - Nikolaev Regional Clinical Hospital, Nikolayev
  - Odessa Regional Hospital, Cardiosurgery Center, Odesa
  - Communal Institution Rivne Regional Clinical Hospital, Rivne
  - Communal Institution of Sumy Regional Rada, Sumy
  - Transcarpathian Regional Clinical Cardiology Clinic, Uzhhorod
  - Communal Institution "Vinnytsia Regional Diagnostic Center of cardiovascular disease", Vinnytsia
  - Vinnytsya Regional Clinical Hospital n.a. Pyrogov, Vinnytsia
  - Zaporizhzhia Regional cardiology dispensary, Zaporizhzhia
- United Kingdom (6):
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - University Hospital of Wales, Cardiff
  - Golden Jubilee Hospital, Clydebank
  - Royal Infirmary of Edinburgh, Edinburgh
  - Altnagelvin Area Hospital, Londonderry
  - Southern Health and Social Care Trust, Portadown

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Goette A, Eckardt L, Valgimigli M, Lewalter T, Laeis P, Reimitz PE, Smolnik R, Zierhut W, Tijssen JG, Vranckx P. Clinical risk predictors in atrial fibrillation patients following successful coronary stenting: ENTRUST-AF PCI sub-analysis. Clin Res Cardiol. 2021 Jun;110(6):831-840. doi: 10.1007/s00392-020-01760-4. Epub 2020 Oct 24. PMID 33098470
- [Derived] Vranckx P, Valgimigli M, Eckardt L, Tijssen J, Lewalter T, Gargiulo G, Batushkin V, Campo G, Lysak Z, Vakaliuk I, Milewski K, Laeis P, Reimitz PE, Smolnik R, Zierhut W, Goette A. Edoxaban-based versus vitamin K antagonist-based antithrombotic regimen after successful coronary stenting in patients with atrial fibrillation (ENTRUST-AF PCI): a randomised, open-label, phase 3b trial. Lancet. 2019 Oct 12;394(10206):1335-1343. doi: 10.1016/S0140-6736(19)31872-0. Epub 2019 Sep 3. PMID 31492505
- [Derived] Vranckx P, Lewalter T, Valgimigli M, Tijssen JG, Reimitz PE, Eckardt L, Lanz HJ, Zierhut W, Smolnik R, Goette A. Evaluation of the safety and efficacy of an edoxaban-based antithrombotic regimen in patients with atrial fibrillation following successful percutaneous coronary intervention (PCI) with stent placement: Rationale and design of the ENTRUST-AF PCI trial. Am Heart J. 2018 Feb;196:105-112. doi: 10.1016/j.ahj.2017.10.009. Epub 2017 Oct 23. PMID 29421002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1506 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study; 1486 participants received treatment. A total of 20 participants (5 Edoxaban and 15 Vitamin K Antagonist) did not receive treatment.
Groups:
- Edoxaban Regimen: Participants who were randomized to Edoxaban 60 mg once-daily or 30 mg once-daily and clopidogrel 75 mg once-daily (or in the presence of a documented clinical need prasugrel [5 mg or 10 mg once-daily] or ticagrelor [90 mg twice-daily] may be used).
- Vitamin K Antagonist Regimen: Participants who were randomized to VKA in combination with clopidogrel 75 mg once-daily (or in the presence of a documented clinical need prasugrel [5 mg or 10 mg once-daily] or ticagrelor [90 mg twice-daily] may be used) and aspirin (100 mg once-daily, for a minimum of 1 month and up to 12 months duration.
Period: Overall Study
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Started | 751 | 755
Completed | 616 | 580
Not Completed | 135 | 175
Not completed — Adverse Event | 56 | 54
Not completed — Withdrawal by Subject | 31 | 52
Not completed — Death | 30 | 23
Not completed — Other | 7 | 14
Not completed — Progressive disease | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 3 | 15
Not completed — Did not receive treatment | 5 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen | Total
Number analyzed (Participants) | 751 | 755 | 1506
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 226 | 202 | 428
  >=65 years | 525 | 553 | 1078
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (9.74) | 70.1 (9.51) | 69.7 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 192 | 386
  Male | 557 | 563 | 1120
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Romania | 17 | 22 | 39
  Hungary | 49 | 54 | 103
  Ukraine | 169 | 175 | 344
  United Kingdom | 6 | 9 | 15
  Portugal | 12 | 12 | 24
  Switzerland | 2 | 5 | 7
  Spain | 58 | 57 | 115
  Austria | 18 | 8 | 26
  Netherlands | 3 | 7 | 10
  South Korea | 50 | 41 | 91
  Belgium | 43 | 37 | 80
  Taiwan | 32 | 46 | 78
  Poland | 74 | 66 | 140
  Italy | 69 | 84 | 153
  France | 21 | 20 | 41
  Lithuania | 24 | 21 | 45
  Serbia | 17 | 11 | 28
  Germany | 87 | 80 | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adjudicated Major or Clinically Relevant Non-major Bleeding As First Event Defined by International Society on Thrombosis and Haemostasis Following Edoxaban-based Regimen Compared With Vitamin K Antagonist (VKA)-Based Regimen
Description: Participants' first major or clinically relevant non-major bleeding (MCRB) events were reported. International Society on Thrombosis and Hemostasis (ISTH) defined bleeding events included: MCRB, major bleeding, including fatal bleeding (intracranial and non-intracranial), symptomatic intracranial hemorrhage, symptomatic bleeding in a critical area or organ, and clinically overt and causing ≥2.0 g/dL adjusted hemoglobin loss, clinically relevant non-major (CRNM) bleeding, minor bleedings, any bleeding (defined as the composite of major, CRNM, and minor bleeding), life-threatening bleeding, provoked (spontaneous, instrumental/traumatic, unknown) bleeding, and spontaneous bleeding.
Time Frame: Day 1 to 12 months postdose
Population: First major or clinically relevant non-major bleeding was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Vitamin K Antagonist Regimen: Participants who were randomized to VKA in combination with clopidogrel 75 mg once-daily (or in the presence of a documented clinical need prasugrel [5 mg or 10 mg once-daily] or ticagrelor [90 mg twice-daily] may be used) and aspirin (100 mg once-daily, for a minimum of 1 month and up to 12 months duration).
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Number analyzed (Participants) | 751 | 755
Participants
  Composite MCRB | 128 | 152
  Major bleeding | 39 | 44
  Clinically relevant non-major bleeding | 89 | 108

2. Secondary Outcome: Number of Participants With Adjudicated Major, Clinically Relevant Non-major and Minor Bleeding (All Events) Defined by International Society on Thrombosis and Haemostasis Following Edoxaban-based Regimen Compared With Vitamin K Antagonist-Based Regimen
Description: All major, clinically relevant non-major and minor bleeding are reported for the secondary outcome. Participants may have experiences more than 1 bleeding event, all occurrences are reported. Participants with International Society on Thrombosis and Hemostasis (ISTH) defined bleeding events included: major or clinically relevant non-major bleeding (MCRB), major bleeding, including fatal bleeding (intracranial and non-intracranial), symptomatic intracranial hemorrhage, symptomatic bleeding in a critical area or organ, and clinically overt and causing ≥2.0 g/dL adjusted hemoglobin loss, clinically relevant non-major (CRNM) bleeding, minor bleedings, any bleeding (defined as the composite of major, CRNM, and minor bleeding), life-threatening bleeding, provoked (spontaneous, instrumental/traumatic, unknown) bleeding, and spontaneous bleeding.
Time Frame: Day 1 to 12 months postdose
Population: All major, clinically relevant non-major, and minor bleeding events were assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Number analyzed (Participants) | 751 | 755
Participants
  Major bleeding | 45 | 48
  Clinically relevant non-major bleeding | 97 | 114
  Minor bleeding | 116 | 125
  Symptomatic intracranial hemorrhage | 4 | 9
  Fatal major bleeding | 1 | 7
  Fatal intracranial hemorrhage | 0 | 4
  Life-threatening bleeding | 5 | 8
  Spontaneous bleeding | 184 | 210

3. Secondary Outcome: Number of Participants With Adjudicated Major, Minor, and Minimal Bleeding by Thrombolysis in Myocardial Infarction (TIMI) Definition Following Edoxaban-based Regimen Compared With Vitamin K Antagonist (VKA)-Based Regimen
Description: Thrombolysis in Myocardial Infarction (TIMI) defined bleeding events included: Major bleeding (including fatal bleeding and non-fatal bleeding [fulfilling the TIMI major bleeding definition], major or minor bleeding, minor bleeding, minimal bleeding, and any bleeding (defined as composite of major, minor, and minimal bleeding)
Time Frame: Day 1 to 12 months postdose
Population: Major, minor, and minimal bleeding was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Number analyzed (Participants) | 751 | 755
Participants
  Major bleeding | 15 | 24
  Fatal bleeding | 1 | 4
  Major or minor bleeding | 124 | 144
  Minor bleeding | 113 | 126
  Minimal bleeding | 117 | 131

4. Secondary Outcome: Number of Participants With Bleeding Academic Research Consortium (BARC) Type 1, 2, 3, and 5 Bleeding According to the BARC Definitions Following Edoxaban-based Regimen Compared With Vitamin K Antagonist (VKA)-Based Regimen
Description: Bleeding Academic Research Consortium (BARC) bleeding events included: Bleeding (defined by BARC type 3 or 5), bleeding (defined by BARC type 2, 3, or 5), and any bleeding (defined as the composite of BARC type 1, 2, 3, or 5), where increases in BARC type indicate worse outcome.
  Type 1: bleeding that is not actionable and does not cause the patient to seek unscheduled performance of studies, hospitalization, or treatment by a healthcare professional; may include episodes leading to self-discontinuation of medical therapy by the patient without consultation; Type 2: any overt, actionable sign of hemorrhage that does not fit the criteria for type 3, 4, or 5 but does meet at least one of the following criteria: (1) requiring nonsurgical, medical intervention, (2) leading to hospitalization or increased level of care, or (3) prompting evaluation; Type 3: Overt bleeding plus hemoglobin drop of 3 to ≤5 g/dL (3a), ≥5 g/dl (3b), and intracranial hemorrhage (3c) Type 5: Fatal bleeding
Time Frame: Day 1 to 12 months postdose
Population: BARC type 1, 2, 3, and 5 bleeding was assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Number analyzed (Participants) | 751 | 755
Participants
  Bleeding (BARC Type 3 or 5) | 36 | 42
  Bleeding (BARC Type 2, 3, or 5) | 124 | 144
  Bleeding (BARC Type 1, 2, 3, or 5) | 207 | 242

5. Secondary Outcome: Number of Participants With Main Efficacy Endpoints For the Overall Study Period Following Edoxaban-based Regimen Compared With Vitamin K Antagonist (VKA)-Based Regimen
Description: The main efficacy endpoints were defined as the composite of cardiovascular death (ARC), stroke (protocol defined), systemic embolic event (SEE), myocardial infarction (MI), or definite stent thrombosis.
Time Frame: Day 1 to 12 months postdose
Population: Efficacy endpoints were assessed in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Number analyzed (Participants) | 751 | 755
Participants
  Composite MEE event | 49 | 46
  Cardiovascular death (ARC) | 10 | 12
  Stroke (Protocol definition) | 10 | 11
  Systemic Embolic Event | 0 | 0
  Myocardial infarction | 22 | 18
  Definite stent thrombosis | 7 | 5

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Following Edoxaban-based Regimen Compared With Vitamin K Antagonist (VKA)-Based Regimen
Description: Treatment-emergent adverse events (TEAEs) in >1.0% of participants were defined as events which started on or after first dose of the assigned study drug (edoxaban and VKA) or started prior to but then worsened after the first dose of the assigned study drug.
Time Frame: Day 1 to 30 days after the last dose
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Number analyzed (Participants) | 746 | 740
Participants
  Any TEAE | 457 | 447
  Infections and Infestations | 145 | 140
  Nasopharyngitis | 25 | 22
  Pneumonia | 20 | 22
  Bronchitis | 19 | 20
  Urinary tract infection | 14 | 19
  Respiratory tract infection | 12 | 15
  Influenza | 10 | 7
  Cardiac Disorders | 136 | 134
  Cardiac failure | 40 | 47
  Atrial fibrillation | 39 | 41
  Bradycardia | 10 | 7
  Cardiac failure congestive | 8 | 8
  Ventricular extrasystoles | 7 | 8
  Tachycardia | 11 | 3
  General Disorders & Administration Site Condition | 113 | 98
  Non-cardiac chest pain | 30 | 24
  Oedema peripheral | 31 | 22
  Asthenia | 21 | 14
  Chest pain | 7 | 11
  Fatigue | 11 | 6
  Gastrointestinal Disorders | 110 | 83
  Diarrhoea | 23 | 19
  Constipation | 11 | 7
  Abdominal pain upper | 6 | 10
  Gastritis | 9 | 5
  Nausea | 8 | 5
  Dyspepsia | 8 | 3
  Respiratory,Thoracic, and Mediastinal Disorders | 87 | 72
  Dyspnoea | 22 | 26
  Cough | 21 | 11
  Dyspnoea exertional | 18 | 5
  Chronic obstructive pulmonary disease | 6 | 10
  Musculoskeletal and Connective Tissue Disorders | 69 | 83
  Back pain | 14 | 14
  Arthralgia | 11 | 12
  Pain in extremity | 5 | 13
  Myalgia | 8 | 8
  Osteoarthritis | 9 | 5
  Investigations | 70 | 79
  Blood creatinine increased | 15 | 13
  Alanine aminotransferase increased | 8 | 13
  Blood pressure increased | 12 | 8
  Creatinine renal clearance decreased | 12 | 7
  Aspartate aminotransferase increased | 7 | 11
  International normalised ratio increased | 0 | 12
  Nervous System Disorders | 83 | 65
  Dizziness | 30 | 22
  Headache | 19 | 12
  Syncope | 8 | 6
  Vascular Disorders | 55 | 62
  Hypertension | 23 | 23
  Hypotension | 14 | 14
  Hypertensive crisis | 11 | 8
  Renal and Urinary Disorders | 49 | 55
  Renal failure | 11 | 12
  Acute kidney injury | 8 | 13
  Renal impairment | 7 | 8
  Injury, Poisoning, and Procedural Complications | 44 | 44
  Fall | 8 | 12
  Skin and Subcutaneous Tissue Disorders | 55 | 33
  Pruritus | 12 | 7
  Rash | 10 | 9
  Metabolism and Nutrition Disorders | 42 | 42
  Gout | 11 | 4
  Blood and Lymphatic System Disorders | 41 | 35
  Anaemia | 19 | 20
  Psychiatric Disorder | 23 | 20
  Insomnia | 8 | 8
  Ear and Labyrinth Disorders | 12 | 16
  Vertigo | 8 | 5

7. Secondary Outcome: Number of Participants With Study Drug-related Treatment-emergent Adverse Events (TEAEs) Experienced by 2 or More Participants Following Edoxaban-based Regimen Compared With Vitamin K Antagonist (VKA)-Based Regimen
Description: Study drug-related treatment-emergent adverse events (TEAEs) (experienced by 2 or more participants) were defined as events which started on or after first dose of the assigned study drug (edoxaban and VKA) or started prior to but then worsened after the first dose of the assigned study drug and were found to be related to treatment by the Investigator.
Time Frame: Day 1 to 30 days after the last dose
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
Number analyzed (Participants) | 746 | 740
Participants
  Any Related TEAE | 57 | 48
  Blood and Lymphatic System Disorders | 12 | 11
  Anaemia | 9 | 7
  Haemorrhagic anaemia | 0 | 2
  Normochromic normocytic anaemia | 2 | 0
  Investigations | 7 | 16
  International normalised ratio increased | 0 | 12
  Blood creatinine increased | 3 | 1
  Creatinine renal clearance decreased | 2 | 2
  Haemoglobin decreased | 2 | 0
  Gastrointestinal Disorders | 12 | 4
  Abdominal pain upper | 3 | 1
  Dyspepsia | 3 | 1
  Nausea | 2 | 0
  Skin and Subcutaneous Tissue Disorders | 6 | 5
  Pruritus | 2 | 1
  Rash | 1 | 2
  Injury, Poisoning, and Procedural Complications | 1 | 7
  Overdose | 0 | 4
  Contusion | 1 | 1
  General Disorders & Administration Site Conditions | 6 | 1
  Death | 3 | 0
  Renal and Urinary Disorders | 2 | 2
  Chronic kidney disease | 1 | 1
  Renal failure | 1 | 1
  Nervous System Disorders | 3 | 0
  Dizziness | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 to 30 days after last dose, up to 2 years, 4 months.
Description: Adverse events were reported from the Safety Analysis Set (746 Edoxaban regimen; 740 Vitamin K Antagonist regimen).
Arm/Group | Edoxaban Regimen | Vitamin K Antagonist Regimen
All-Cause Mortality (participants affected / at risk) | 46/746 | 37/740
Serious Adverse Events (participants affected / at risk) | 176/746 | 175/740
Other Adverse Events (participants affected / at risk) | 457/746 | 447/740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban Regimen (N=746) | Vitamin K Antagonist Regimen (N=740)
Cardiac failure (Cardiac disorders) | 29 | 35
Atrial fibrillation (Cardiac disorders) | 20 | 14
Pneumonia (Infections and infestations) | 14 | 13
Urinary tract infection (Infections and infestations) | 3 | 2
Cellulitis (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 3 | 1
Appendicitis (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Aeromonas infection (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Device-related infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peritoneal abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Amyloidosis (Immune system disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 0
Sciatica (Nervous system disorders) | 1 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cervicogenic headache (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 6 | 5
Cardiac failure acute (Cardiac disorders) | 2 | 4
Sinus node dysfunction (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 3 | 1
Cardiac failure chronic (Cardiac disorders) | 3 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 3
Aortic valve stenosis (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 3 | 0
Atrial tachycardia (Cardiac disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 2
Aortic dissection (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Dental cyst (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 4
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Biliary fistula (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 7
Renal failure (Renal and urinary disorders) | 5 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Spermatocele (Reproductive system and breast disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 6 | 3
Death (General disorders) | 4 | 3
Sudden death (General disorders) | 1 | 3
Chest pain (General disorders) | 2 | 1
Vascular stent thrombosis (General disorders) | 2 | 1
Asthenia (General disorders) | 2 | 0
Vascular stent restenosis (General disorders) | 2 | 0
Chest discomfort (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Costal cartilage fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Product use issue (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 0 | 1
Device capturing issue (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban Regimen (N=746) | Vitamin K Antagonist Regimen (N=740)
Nasopharyngitis (Infections and infestations) | 25 | 22
Pneumonia (Infections and infestations) | 20 | 22
Bronchitis (Infections and infestations) | 19 | 20
Urinary tract infection (Infections and infestations) | 14 | 19
Respiratory tract infection (Infections and infestations) | 12 | 15
Influenza (Infections and infestations) | 10 | 7
Cardiac failure (Cardiac disorders) | 40 | 47
Atrial fibrillation (Cardiac disorders) | 39 | 41
Bradycardia (Cardiac disorders) | 10 | 7
Cardiac failure congestive (Cardiac disorders) | 8 | 8
Ventricular extrasystoles (Cardiac disorders) | 7 | 8
Tachycardia (Cardiac disorders) | 11 | 3
Non-cardiac chest pain (General disorders) | 30 | 24
Oedema peripheral (General disorders) | 31 | 22
Asthenia (General disorders) | 21 | 14
Chest pain (General disorders) | 7 | 11
Fatigue (General disorders) | 11 | 6
Diarrhoea (Gastrointestinal disorders) | 23 | 19
Constipation (Gastrointestinal disorders) | 11 | 7
Abdominal pain upper (Gastrointestinal disorders) | 6 | 10
Gastritis (Gastrointestinal disorders) | 9 | 5
Nausea (Gastrointestinal disorders) | 8 | 5
Dyspepsia (Gastrointestinal disorders) | 8 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 18 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 5
Blood creatinine increased (Investigations) | 15 | 13
Alanine aminotransferase increased (Investigations) | 8 | 13
Blood pressure increased (Investigations) | 12 | 8
Creatinine renal clearance increased (Investigations) | 12 | 7
Aspartate aminotransferase increased (Investigations) | 7 | 11
International normalised ratio increased (Investigations) | 0 | 12
Dizziness (Nervous system disorders) | 30 | 22
Headache (Nervous system disorders) | 19 | 12
Syncope (Nervous system disorders) | 8 | 6
Hypertension (Vascular disorders) | 23 | 23
Hypotension (Vascular disorders) | 14 | 14
Hypertensive crisis (Vascular disorders) | 11 | 8
Renal failure (Renal and urinary disorders) | 11 | 12
Acute kidney injury (Renal and urinary disorders) | 8 | 13
Renal impairment (Renal and urinary disorders) | 7 | 8
Fall (Injury, poisoning and procedural complications) | 8 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 7
Rash (Skin and subcutaneous tissue disorders) | 10 | 9
Gout (Metabolism and nutrition disorders) | 11 | 4
Anaemia (Blood and lymphatic system disorders) | 19 | 20
Insomnia (Psychiatric disorders) | 8 | 8
Vertigo (Ear and labyrinth disorders) | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT02866175/Prot_SAP_000.pdf